CLINICAL TRIAL: NCT03024502
Title: Randomized Clinical Trial of a Mucoadhesive Gel Containing EPP-AF in Patients Diagnosed With Vulvovaginal Candidiasis
Brief Title: Patients With Vulvovaginal Candidiasis
Acronym: EPP-AFG-VVC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Silvana Maria Quintana, clinical professor and principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03.12.0056.00; 2013/50496-2 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Vulvovaginal Candidiasis
Keywords: vulvovaginal candidiasis; EPPAF mucoadhesive gel; clotrimazol
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Clotrimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EPP-AF Gel 1% (Experimental): Group of patients that will be treated with EPP-AF mucoadhesive gel 1%, during 7 day, 1x/day.
  Interventions: Drug: EPP-AF Gel 1%
- Clotrimazole cream (Experimental): Group of patients that will be treated with clotrimazole cream, during 7 day, 1x/day.
  Interventions: Drug: Clotrimazole
- EPP-AF Gel 2% (Experimental): Group of patients that will be treated with EPP-AF mucoadhesive gel 2%, during 7 day, 1x/day.
  Interventions: Drug: EPP-AF Gel 2%

INTERVENTIONS:
Drug: EPP-AF Gel 1% — Administration intravaginal of EPP-AG Gel 1%, 1x/day, 7 days
  Other Names: Drug 1
  Arms: EPP-AF Gel 1%
Drug: EPP-AF Gel 2% — Administration intravaginal of EPP-AG Gel 1%, 1x/day, 7 days
  Other Names: Drug 2
  Arms: EPP-AF Gel 2%
Drug: Clotrimazole — Administration intravaginal of clotrimazol, 1x/day, 7 days
  Other Names: Active Comparator
  Arms: Clotrimazole cream

SUMMARY:
The present study aims to evaluate the safety of two mucoadhesive gels containing a propolis standardized extract identified as EPP-AF, with 1 and 2% of propolis. The efficacy studies with both propolis gels will be performed in comparison with clotrimazole cream in patients presenting vulvovaginal candidiasis.

DETAILED DESCRIPTION:
Vaginal candidiasis is the second infection of the genital tract after bacterial vaginosis. Up to 75% of women will have at least one episode in their lives, but the clinical manifestations can be very variable. Around 10 to 20% will be asymptomatic and 5 to 10% will have the recurrent candidiasis that means 4 or more episodes in a year. The predominant symptoms are pruritus in 89% and burning during urination and sexual intercourse in 66%. The therapeutic regimen for acute fungal infections by C. albicans should consider the intensity of the clinical symptoms, recurrence, patient preference for the route of administration and consequent adherence to treatment, presence of pregnancy and the possibility of side effects. In general, the schemes include anti-fungal substances of the azoles type. Intravaginal administration of drugs requires the development of formulations suited to the area and adherence to the treatment can be increased if mucoadhesive formulations are obtained which avoid discomfort and provide adequate release of the active compounds. In this sense, the present project had the objective of developing a mucoadhesive gel containing Propolis Standardized (EPP-AF®) for the treatment of vaginal candidiasis, especially since preclinical efficacy and safety data demonstrated the clinical potential of the product. So the present proposal aims at the clinical study evaluate the efficacy of two formulations with 1 and 2% of propolis in comparison with clotrimazole cream treatment (patients affected by Candidiasis) and also evaluate the safety of both propolis gels in healthy volunteers. The efficacy protocol of the test product in patients with vaginal candidiasis will be performed in an open-label, randomized, three-arm, clinical trial with active clotrimazole-based control. Patients will be recruited (T0) and evaluated at 10 and 30 days after initiation of treatment, and the primary outcome will be the clinical cure rate.

ELIGIBILITY:
Inclusion Criteria:

-Have performed the clinical and laboratory diagnosis of vulvovaginitis by Candida

Exclusion Criteria:

* cPatients with recurrent candidiasis;
* History of hepatic, renal, hematological, cardiovascular diseases and with decompensated diabetes mellitus (glycemia above 200) and obesity with BMI above 35);
* Diagnosis of vulvovaginitis by another agent;
* Make use of chronic antimicrobials (informed by the patient)
* Be pregnant
* Allergy to some component of medications given

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
clinical cure | 10 days
  Participants will be evaluated on the tenth day after insertion in the study (on the third day after the termination of the vaginal cream). The clinical cure will be evaluated by means of a questionnaire and specular examination. The possibilities will be:
  1. Candidacy Resolution
  2. No resolution of candidiasis
  The questionnaire will be:
  Pruritus: yes or no Burning: yes or no Dysuria: yes or no Edema of the genital area: yes or no Running: yes or no
  The specular examination will evaluate:
  Presence of hyperemia: yes or no Edema of the genital area: yes or no Presence of cracks: yes or no Pathological vaginal contents: yes or no The positive response to any of the questions or signs / symptoms will be considered as clinical failure

SECONDARY OUTCOMES:
microbiology cure | 10 days
  Participants will be evaluated on the tenth day after insertion in the study (on the third day after the termination of the vaginal cream). The patient's clinical complaint will be evaluated and the specular examination will be performed. In this evaluation will be collected the following exams:
  Vaginal pH measurement:
  Normal 3.5 to 4.5 Abnormal> 4.5
  Bacterioscopy with KOH10%:
  Normal: absence of pseudohifas or other pathogenic elements Abnormal: presence of pseudohifas
  Culture for candida albicans:
  Normal: Negative Abnormal: positive
  PCR for candida:
  Normal negative Abnormal: positive
  The possibilities will be:
  1. Candidacy Resolution
  2. No resolution of candidiasis It will be considered microbiological cure when all laboratory tests are considered normal

CONTACTS AND LOCATIONS:
Overall Officials: silvana m quintana, phd, Principal Investigator — Sao Paulo University
Locations (1):
- Clinical Hospital of Sao Paulo University, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No